CLINICAL TRIAL: NCT06553482
Title: Impact of Exercise Training at Maximal Fat Oxidation (FatMax) Intensity on Metabolic and Epigenetic Parameters in Subjects With Excessive Body Mass: Study Protocol of a Randomized Controlled Trial
Brief Title: FatMax Training on Metabolic and Epigenetic Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Marco Antonio Hernández Lepe, Principal Investigator, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LNC-2023-69
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity; Body Weight Changes
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: The subjects assigned to each group will participate in a randomized clinical trial, with a duration of 16 weeks of intervention. Measurements of all variables will be taken on the first day of the evaluation (considered the basal state) and at the end of 16 weeks of the intervention according to the group in which they were randomized, to be followed by sta-tistical analysis of the data. The variables contemplated involve assessments of body composition and physical capacities, biochemical variables, epigenetic variables and alternate variables.
Who Masked: Outcomes Assessor
Masking Description: Statistical Analysis will be conducted without knowledge of gropus allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FatMax group (Experimental): low-intensity exercise training sessions (FatMax zone)
  Interventions: Other: FatMAx training intervention
- FatMAx and musuclar endurance exercise group (Experimental): FatMax zone exercises as well as muscular resistance exercises
  Interventions: Other: FatMax and physical endurance exercise intervention
- Control (Active Comparator): Group without physical activity intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: FatMAx training intervention — FatMax training program on a treadmill or stationary bicycle, whichever is more convenient for them
  Arms: FatMax group
Other: FatMax and physical endurance exercise intervention — FatMax training program on a treadmill or stationary bicycle, whichever is more convenient for them, with muscular endurance exercise
  Arms: FatMAx and musuclar endurance exercise group
Other: Control — No intervention pf physical activity
  Arms: Control

SUMMARY:
Exercise is an essential pillar for the health of all individuals, as it contributes to physical, mental, and emotional well-being. Various international organizations, such as the World Health Organization, advocate for the integration of exercise into healthy lifestyles, recognizing its im-portance in disease prevention and improving quality of life. However, despite the general consensus on its value, there is no universal agreement on specific prescriptions for vulnerable groups, highlighting the need for personalized approaches that consider the unique characteristics and needs of each individual. It has been proposed that a moderate aerobic exercise training program could promote positive outcomes in individuals living with overweight and obesity, particularly with an emphasis on reducing injury risk, ensuring high adherence, and achieving favorable health changes. In this regard, the present protocol establishes the basis for a randomized clinical trial based on exercise prescription at the maximal fat oxidation rate in young individuals with overweight and obesity, with a duration of 16 weeks. Throughout the study, biochemical changes (cholesterol, glucose, triglycerides, and inflammatory markers), metabolic changes (de-termination of fat and carbohydrate utilization rates during rest and exercise), and epigenetic changes (focusing on microRNAs associated with adipogenesis, inflammation, and fat metabolism) will be monitored.

DETAILED DESCRIPTION:
Obesity is a public health problem that affects millions of people in Mexico and around the world. This disease has not only increased alarmingly in recent decades but has also been recognized as one of the main risk factors for chronic diseases such as dia-betes, cardiovascular disease, and certain types of cancer. By 2022, it was estimated that 890 million adults were living with obesity and the trend continues to in-crease with obesity occurring at younger and younger ages.

The critical levels of this disease urgently demand the need to address this crisis on multiple fronts. Traditional strategies to combat obesity have focused primarily on individual responsibility, emphasizing the need to improve diet and increase physical activity. However, reducing obesity to a mere problem of willpower is insufficient to under-stand the complexity of the problem, which involves genetic, psychological, social, eco-nomic, environmental and, above all, individual factors, where dietary and exercise pre-scription is fundamental for its efficacy and adherence by those affected.

In this sense, it is crucial to conduct studies that explore the effectiveness of training and physical activity programs specifically designed for people with obesity. These pro-grams should not only focus on improving biological markers of health, such as body fat reduction, lipid profile improvement, maintenance of lean mass or exercise-associated injury limitations, but also on promoting long-term adherence and the creation of healthy habits. Understanding how to adapt exercise to the specific needs of this population is essential to develop more effective and sustainable interventions.

If these issues are not specifically addressed, the consequences will be serious. The prevalence of obesity will continue to rise, increasing the number of people at risk of de-veloping chronic diseases, reducing their life expectancy and quality of life. In addition, the health care system will face increased costs and pressure, which will make this silent pandemic even more difficult to manage. Thus, the present protocol aims to evaluate the effect of a personalized physical training program at maximum fat oxidation (FatMax) for 16 weeks on biochemical, metabolic and epigenetic parameters in overweight and obese young adults.

The subjects assigned to each group will participate in a randomized clinical trial, with a duration of 16 weeks of intervention. Measurements of all variables will be taken on the first day of the evaluation (considered the basal state) and at the end of 16 weeks of the intervention according to the group in which they were randomized, to be followed by sta-tistical analysis of the data. The variables contemplated involve assessments of body composition and physical capacities, biochemical variables, epigenetic variables and alternate variables.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Daily energy expenditure <4 METs
* Body mass index ≥25 kg/m2
* Acceptance of informed consent

Exclusion/elimination Criteria:

* ≥100 ml of alcohol consumption per week
* Consume a dietary supplement or pharmacological treatment
* Have limitations to perform regular physical activity
* Have a chronic non-communicable disease
* Answer "yes" to any of the questions on the Physical Activity Readiness- Questionnaire for Everyone (PAR-Q+); which represents a health risk.
* <80% attendance at exercise sessions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Body composition change | 16 weeks
  Changes in body composition (fat mass and muscle mass) after the intervention

SECONDARY OUTCOMES:
Changes in lipid profile | 16 weeks
  Changes in total cholesterol, high-density lipoprotein cholesterol (c-HDL), low-density lipoprotein cholesterol (c-LDL), triglycerides
Changes in epigenetic markers | 16 weeks
  Changes in microRNAs involved in inflammatory processes (miR-15, miR-29c, miR-30a, miR-142/3, miR-181a), adipogenesis (miR-188-5p, miR-146b-5p, miR-103, miR-107, miR-125b), and fatty acid metabolism (miR-33, miR-335, miR-370, miR-758)

CONTACTS AND LOCATIONS:
Overall Officials: René Bassó-Quevedo, MSc, Study Chair — Bioethic Comittee of the Autonomous University of Baja California
Locations (1):
- Medical and Psychology School, Tijuana, California, Mexico

IPD SHARING:
Plan to Share IPD: No
Publication of manuscripts without any name of a participant

REFERENCES:
- [Background] Chavez-Guevara IA, Urquidez-Romero R, Perez-Leon JA, Gonzalez-Rodriguez E, Moreno-Brito V, Ramos-Jimenez A. Chronic Effect of Fatmax Training on Body Weight, Fat Mass, and Cardiorespiratory Fitness in Obese Subjects: A Meta-Analysis of Randomized Clinical Trials. Int J Environ Res Public Health. 2020 Oct 28;17(21):7888. doi: 10.3390/ijerph17217888. PMID 33126461
- [Background] Brun JF, Myzia J, Varlet-Marie E, Raynaud de Mauverger E, Mercier J. Beyond the Calorie Paradigm: Taking into Account in Practice the Balance of Fat and Carbohydrate Oxidation during Exercise? Nutrients. 2022 Apr 12;14(8):1605. doi: 10.3390/nu14081605. PMID 35458167
- [Background] Pico-Sirvent I, Manresa-Rocamora A, Aracil-Marco A, Moya-Ramon M. A Combination of Aerobic Exercise at Fatmax and Low Resistance Training Increases Fat Oxidation and Maintains Muscle Mass, in Women Waiting for Bariatric Surgery. Obes Surg. 2022 Apr;32(4):1130-1140. doi: 10.1007/s11695-022-05897-1. Epub 2022 Jan 20. PMID 35048250
- [Background] Chavez-Guevara IA, Amaro-Gahete FJ, Ramos-Jimenez A, Brun JF. Toward Exercise Guidelines for Optimizing Fat Oxidation During Exercise in Obesity: A Systematic Review and Meta-Regression. Sports Med. 2023 Dec;53(12):2399-2416. doi: 10.1007/s40279-023-01897-y. Epub 2023 Aug 16. PMID 37584843
- [Background] Wang D, Zhang P, Li J. Crossover point and maximal fat oxidation training effects on blood lipid metabolism in young overweight women: a pilot study. Front Physiol. 2023 Jun 16;14:1190109. doi: 10.3389/fphys.2023.1190109. eCollection 2023. PMID 37398909
- [Derived] Hernandez-Lepe MA, Hernandez-Ontiveros DA, Chavez-Guevara IA, Ramos-Jimenez A, Hernandez-Torres RP, Lopez-Fregoso RJ, Ramos-Lopez O, Amaro-Gahete FJ, Muniz-Salazar R, Olivas-Aguirre FJ. Impact of Exercise Training at Maximal Fat Oxidation Intensity on Metabolic and Epigenetic Parameters in Patients with Overweight and Obesity: Study Protocol of a Randomized Controlled Trial. J Funct Morphol Kinesiol. 2024 Oct 31;9(4):214. doi: 10.3390/jfmk9040214. PMID 39584867